CLINICAL TRIAL: NCT00229190
Title: Reproducibility of Cell Counts in Nasal Lavage: A Comparison of Pooled Versus Non-Pooled Nasal Lavage Samples
Brief Title: Nasal Lavage Study: Comparing Single Versus Multi Sample Lavages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Firestone Institute for Respiratory Health (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-227; 2003/11
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Nasal Lavage Fluid; Eosinophils; Reproducibility of Results
Keywords: Nasal lavage fluid; Eosinophils; Reproducibility of results
MeSH Terms: interventions — Nasal Lavage; Skin Tests; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Nasal lavage
Procedure: Allergy skin testing
Procedure: Peak nasal inspiratory flow
Procedure: Acoustic rhinometry
Procedure: Nasal examination
Procedure: Quality of Life Questionnaire
Procedure: Physical examination

SUMMARY:
Nasal lavage could be an integral component of assessing airway inflammation. Research into the reproducibility of cell counts is key to understanding the value of lavage results.

The objective of this study is to evaluate and compare the reproducibility of a common nasal lavage technique and its variation in a sample of subjects with nasal symptoms (e.g. runny nose, congestion, sneezing, post nasal drip), and in individuals without nasal symptoms.

DETAILED DESCRIPTION:
Nasal lavage is a relatively simple way to measure the degree of upper airway inflammation. It is useful in research because it is noninvasive, relatively discomfort-free, and simple to perform. Yet there is no standardized method for collecting upper airway cells. The definition of nasal lavage can differ widely between research groups. The method, and its pooled modification, chosen for this trial are based on the commonly used Naclerio technique.

Upper airway inflammation is linked to a broad spectrum of disease: nasal polyposis, seasonal and perennial allergic rhinitis, vasomotor or non-allergic rhinitis, and sinusitis. Assessing the degree of upper airway inflammation through objective measures has obvious clinical and research benefits. For example, nasal polyps contain a large number of activated eosinophils - about 20% of the constituents of nasal polyp tissue. Allergic rhinitis is also associated with elevated inflammatory cell counts - eosinophils, basophils, mast cells, lymphocytes and their mediators. The impact of treatment on nasal inflammation is a key factor in the evaluation of new nasal polyp or allergic rhinitis therapies. Therefore it is imperative that nasal inflammation measurements be evaluated for reliability.

As nasal inflammation is present in a variety of diseases, a cross section of subjects will be enrolled in this trial. Nasal lavages will be performed on nasal polyp subjects, perennial allergic rhinitis subjects, and normal subjects. This project will assess the repeatability of a single sample lavage in comparison to the repeatability of a modified version, i.e. a lavage sample conducted three times, 15 minutes apart, and then pooled, or combined. We expect to find the highest eosinophil counts in patients with nasal polyposis, intermediate levels in patients with perennial allergic rhinitis and low levels in normal subjects, based on previous work.

This project will be a single-centre, randomized trial involving three sets of seven subjects - polyp subjects, perennial allergic rhinitis subjects, and normals. All subjects will be blinded to the assessment of outcome measurements.

The study will be comprised of four clinic appointments. Appointments will be scheduled seven to 10 days apart. All subjects will be randomly assigned their lavage sampling group at their baseline visit. Group one will consist of a single sample lavage at visit one, a multiple sample lavage at visit two, a single sample lavage at visit three, and a multiple sample lavage a visit four. Group two will be the reverse order.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged 18 years or older.
* Subject understands the research project and agrees to participate by signing an informed consent agreement.
* Subject is able to successfully complete nasal lavage training session.

Exclusion Criteria:

* Subjects with severe nasal polyps which prevent collecting adequate nasal lavage sample.
* Subjects who have undergone surgery to treat their nasal polyps (nasal polypectomy) within one year prior to visit one
* Subjects who have a known fungal infection of the nose and/or paranasal sinuses, nasal candidiasis, acute or chronic infectious sinusitis of viral or bacterial nature.
* Subjects who have had an upper respiratory tract infection within four weeks prior to visit one.
* Subjects having cystic fibrosis, Young's syndrome, primary ciliary dyskinesia, known HIV infection or alcohol abuse.
* Subjects with clinically significant, uncontrolled evidence of cardiovascular, neurological, hepatic, renal, respiratory, or any other medical condition that may interfere with the study.
* Subjects with a recent history (within six months) of a clinically significant psychiatric disorder other than mild depression.
* Subjects who have any clinically relevant deviation from normal in the general physical examination.
* Subjects who have received any depot, systemic or oral corticosteroid in the previous three months prior to the start of the study.
* Subjects who are using an intranasal steroid or antihistamine for their nasal symptoms and are unable to remain on a constant dose for four weeks prior to visit 1 or for the duration of the study.
* Females who are pregnant or lactating or are likely to become pregnant during the study or are less than 8 weeks postpartum. Women of childbearing age may be included if, in the opinion of the investigator, they are taking adequate contraceptive measures.
* Subjects who are unable to follow the instructions within this protocol or known inability to attend all clinic visits within the intervals stated.
* Subjects who have participated in a clinical trial involving an investigational or marketed drug within four weeks of visit one.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21
Dates: Start 2004-09; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Eosinophil per cent of cells recovered in lavage fluid

SECONDARY OUTCOMES:
Albumen concentration in lavage fluid

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keith, MD MSc FRCPC, Principal Investigator — Hamilton Health Sciences Corporation, McMaster Site
Locations (1):
- Hamilton Health Sciences Corporation, McMaster Site, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Naclerio RM, Meier HL, Kagey-Sobotka A, Adkinson NF Jr, Meyers DA, Norman PS, Lichtenstein LM. Mediator release after nasal airway challenge with allergen. Am Rev Respir Dis. 1983 Oct;128(4):597-602. doi: 10.1164/arrd.1983.128.4.597. PMID 6354022
- [Background] Finotto S, Dolovich J, Denburg JA, Jordana M, Marshall JS. Functional heterogeneity of mast cells isolated from different microenvironments within nasal polyp tissue. Clin Exp Immunol. 1994 Feb;95(2):343-50. doi: 10.1111/j.1365-2249.1994.tb06535.x. PMID 7508349
- [Background] Koren HS, Hatch GE, Graham DE. Nasal lavage as a tool in assessing acute inflammation in response to inhaled pollutants. Toxicology. 1990 Jan-Feb;60(1-2):15-25. doi: 10.1016/0300-483x(90)90159-e. PMID 2315937
- [Background] Miadonna A, Milazzo N, Gibelli S, Salmaso C, Lorini M, Tedeschi A. Nasal response to a single antigen challenge in patients with allergic rhinitis - inflammatory cell recruitment persists up to 48 hours. Clin Exp Allergy. 1999 Jul;29(7):941-9. doi: 10.1046/j.1365-2222.1999.00609.x. PMID 10383595
- [Background] Noah TL, Henderson FW, Henry MM, Peden DB, Devlin RB. Nasal lavage cytokines in normal, allergic, and asthmatic school-age children. Am J Respir Crit Care Med. 1995 Oct;152(4 Pt 1):1290-6. doi: 10.1164/ajrccm.152.4.7551384.
- [Background] Nikasinovic-Fournier L, Just J, Seta N, Callais F, Sahraoui F, Grimfeld A, Momas I. Nasal lavage as a tool for the assessment of upper-airway inflammation in adults and children. J Lab Clin Med. 2002 Mar;139(3):173-80. doi: 10.1067/mlc.2002.121661. PMID 11944028
- [Background] Belda J, Parameswaran K, Keith PK, Hargreave FE. Repeatability and validity of cell and fluid-phase measurements in nasal fluid: a comparison of two methods of nasal lavage. Clin Exp Allergy. 2001 Jul;31(7):1111-5. doi: 10.1046/j.1365-2222.2001.01133.x. PMID 11468003
- [Background] Greiff L, Pipkorn U, Alkner U, Persson CG. The 'nasal pool' device applies controlled concentrations of solutes on human nasal airway mucosa and samples its surface exudations/secretions. Clin Exp Allergy. 1990 May;20(3):253-9. doi: 10.1111/j.1365-2222.1990.tb02680.x. PMID 2364306
- [Background] Hauser R, Garcia-Closas M, Kelsey KT, Christiani DC. Variability of nasal lavage polymorphonuclear leukocyte counts in unexposed subjects: its potential utility for epidemiology. Arch Environ Health. 1994 Jul-Aug;49(4):267-72. doi: 10.1080/00039896.1994.9937478. PMID 8031183
- [Background] Sulakvelidze I, Conway M, Evans S, Stetsko PI, Djuric V, Dolovich J. Clinical and nasal irrigation fluid findings in perennial allergic rhinitis. Am J Rhinol. 1997 Nov-Dec;11(6):435-41. doi: 10.2500/105065897780914965. PMID 9438056
- [Background] Keith PK, Conway M, Evans S, Wong DA, Jordana G, Pengelly D, Dolovich J. Nasal polyps: effects of seasonal allergen exposure. J Allergy Clin Immunol. 1994 Mar;93(3):567-74. doi: 10.1016/s0091-6749(94)70068-0. PMID 8151059
- [Background] Austin CE, Foreman JC. Acoustic rhinometry compared with posterior rhinomanometry in the measurement of histamine- and bradykinin-induced changes in nasal airway patency. Br J Clin Pharmacol. 1994 Jan;37(1):33-7. doi: 10.1111/j.1365-2125.1994.tb04235.x. PMID 8148216
- [Background] Juniper EF. Measuring health-related quality of life in rhinitis. J Allergy Clin Immunol. 1997 Feb;99(2):S742-9. doi: 10.1016/s0091-6749(97)90000-2. PMID 9042066
- [Background] Keith PK, Conway M, Dolovich J.Development and validation of a nasal-polyposis quality of life questionniare. Journal of Allergy and Clinical Immunology 1996;97:192 (Abstract)